CLINICAL TRIAL: NCT03612037
Title: Impact of Alpha-Lipoic Acid Ingestion on Glucose Tolerance in Subjects With Pre-Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Todd Rideout, Associate Professor, State University of New York at Buffalo
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MODCR00002022
Record Dates: First submitted 2018-07-16; First posted 2018-08-02 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: PreDiabetes
Keywords: pre-diabetes; glucose; insulin; blood lipids; alpha lipoic acid
MeSH Terms: conditions — Prediabetic State; Glucose Intolerance; Insulin Resistance | interventions — Thioctic Acid; Cellulose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Phase (Placebo Comparator): cellulose (600 mg)
  Interventions: Dietary Supplement: Cellulose
- Experimental Phase (Experimental): alpha lipoic acid (600 mg)
  Interventions: Dietary Supplement: alpha lipoic acid

INTERVENTIONS:
Dietary Supplement: alpha lipoic acid — 600 mg/day oral dose of alpha lipoic acid
  Arms: Experimental Phase
Dietary Supplement: Cellulose — 600mg/day oral dose of placebo cellulose
  Arms: Control Phase

SUMMARY:
Obesity, with a prevalence of over 35% in American adults, is considered the most critical threat to the health and well-being of Americans. Obesity-associated metabolic abnormalities, including hyperglycemia, insulin resistance, and dyslipidemia, contribute substantially to elevated risk of cardiovascular disease (CVD) and diabetes. Although significant and sustained lifestyle modifications in diet and exercise are effective in reducing weight and improving obesity-related metabolic disturbances, long-term compliance to drastic changes in diet and daily activity patterns is often difficult to attain given the hectic lifestyle of modern societies. Health-promoting nutraceuticals - naturally occurring bioactive compounds capable of eliciting targeted molecular responses at the cellular level - may be an effective and convenient strategy to assist in weight reduction and reduce disease risk factors in obese individuals. Furthermore, nutraceutical compounds could prove to be a powerful adjunct to lifestyle and pharmacological weight reduction therapies, as they are relatively safe, cost effective, and possess the ability to modulate specific, and sometimes multiple, molecular targets. As a dietary supplement, alpha-lipoic acid appears to have broad molecular specificity with an impressive array of metabolic health benefits that include weight loss, reduction in blood lipids, and improved glycemic control. As the effects of alpha-lipoic acid supplementation for dyslipidemia, hyperglycemia, and body composition through appetite suppression and increased energy expenditure have been repeatedly confirmed in multiple animal models, it is surprising that there has been limited effort to translate these responses to human subjects. Given the strong pre-clinical data supporting the health benefits of alpha-lipoic acid, there is a clear need to conduct controlled interventions to address the current clinical knowledge gap and assess if the anti-diabetic effect of α-lipoic acid can be translated to humans.

The primary objective of this application is to determine the efficacy of alpha-lipoic acid supplementation on glycemic control and body composition in obese pre-diabetic adults. The investigators hypothesize that alpha-lipoic acid supplementation will improve biomarkers of diabetes and cardiovascular risk and promote changes in body composition in obese adults.

ELIGIBILITY:
Inclusion Criteria:

* sedentary individuals (exercises < 2 days/week)
* fasting blood glucose between 100-125 mg/dl (pre-diabetes)
* BMI of 25-40.

Exclusion Criteria:

* physically active lifestyle (exercise > two days/week)
* pregnancy
* history of cigarette smoking
* medication and/or dietary supplement to control blood glucose, lipids, or blood pressure.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Glycemic control | 1 month
  blood glucose and insulin

SECONDARY OUTCOMES:
Blood lipids | 1 month
  Blood cholesterol
Blood lipids | 1 month
  Triglycerides

IPD SHARING:
Plan to Share IPD: No